CLINICAL TRIAL: NCT06233786
Title: Effectiveness of Non-invasive Neuromodulation in Primary Dysmenhorrea: A Randomized Clinical Trial
Brief Title: The Effectivenes of Non-invasive Neuromodulation in Adult Women With Primary Dysmenorrhea, Through the TENS Stimulation at Different Times of Mentrual Cycle in Each Group
Acronym: Dysmenorrhea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naiara Benítez Aramburu (Other)
Responsible Party: Sponsor-Investigator, Naiara Benítez Aramburu, Principal investigator, Escoles Universitaries Gimbernat
Organization: Escoles Universitaries Gimbernat (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.211
Record Dates: First submitted 2024-01-11; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Transcutaneous Electrical Nerve Stimulation; Non-Invasive Neuromodulation; Sacral Surface Stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS in the bleeding phase (Experimental): After completing the screening questionnaire and being evaluated, they receive TENS stimulation in the menstrual phase between days 25-28 (days before bleeding and where symptoms may begin) and 1-3 (first days of bleeding). They are evaluated again immediately after treatment and at the beginning of the next bleeding phase, being 28 days after the intervention.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- TENS in the luteal phase (Experimental): After completing the screening questionnaire and being evaluated, they receive TENS stimulation TENS stimulation in the luteal phase between days 17 to 24 of the menstrual cycle after the start of bleeding. They are evaluated again at the beginning of the next bleeding phase, being 7 days after the intervention, as well as 28 days after, being the next cycle.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Sham TENS in the bleeding phase (Sham Comparator): Same procedure as TENS in the bleeding phase, but without TENS stimulation.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — This intervention is performed using a TENS with an asymmetric biphasic wave of 200 µs width, frequency of 100Hz and maximum intensity tolerated by the participant, adapting to avoid accommodation. The intervention will be carried out for 30 minutes, once a day, and 2 days a week, with 48-72 hours between both interventions. Regarding the electrodes, 4 adhesive electrodes (5.0x5.0) will be placed, 2 in the lower lumbar region and two in the parasacral region (S2-S4).

SUMMARY:
The effectiveness of non-invasive neuromodulation in adult women with primary dysmenorrhea, through the TENS stimulation at different times in each group: during the bleeding phase (G1), between days 25-28 and 1-3 of menstrual cycle, and in the luteal phase (GI2), between days 17 to 24 of menstrual cycle.

The control group (CG) will be treated just like GI1, during the bleeding phase, but without the TENS transmitting the current. Participants will be evaluated by the NPRS, MPQ, SF12, CVM-22, HADS, PCS, PSQI and UDP immediately after treatment in GI1 and GC, and at the beginning of the next bleeding phase, being 28 days after the intervention in the case of GI1 and GC, and 7 days after the intervention in the case of GI2, as well as 28 days after in this last.

DETAILED DESCRIPTION:
This RCT evaluates women of legal age, with pain greater than 3 on the NPRS scale, and whose menstrual cycle is regular, considered regular between 25-30 days. The sample will be divided into a cases group which in turn will be divided into 2 subgroups: stimulation intervention in women with dysmenorrhea during the bleeding phase (GI1), and in the luteal phase (GI2). On the other hand, the control group (CG) will be treated just like GI1, during the bleeding phase, but without the transcutaneous electrical nerve stimulation (TENS) transmitting the current.

Initially, a screening questionnaire will be completed. Subsequently, a first assessment will be done to all included participants, which will be conducted by completing the Numerical Pain Scale (NPRS) in relation to their pain for 5 days, McGill Pain Questionnaire (MPQ), SF12 Health Survey, Specific Quality of life Questionnaire Related to Menstruation (CVM-22), Hospital Anxiety and Depression Scale (HADS) and Pain Catastrophizing Scale (PCS) and Pittsburgh Sleep Quality Index (PSQI), as well as pressure pain threshold measure (PPT). Participants will also be evaluated immediately after treatment and at the beginning of the next bleeding phase (next menstrual cycle), being 28 days after the intervention in the case of GI1 and GC, and 7 days after the intervention in the case of GI2.

Regarding the intervention, the treatment plan to be done will be as follows:

* GI1: TENS stimulation in the menstrual phase between days 25-28 (days before bleeding and where symptoms may begin) and 1-3 (first days of bleeding).
* GI2: TENS stimulation in the follicular phase between days 17 to 24 of the menstrual cycle after the start of bleeding.
* GC: Same procedure as GI1, but without TENS stimulation.

This intervention is performed using a TENS with an asymmetric biphasic wave of 200 µs width, frequency of 100Hz and maximum intensity tolerated by the participant, adapting to avoid accommodation. The intervention will be carried out for 30 minutes, once a day, and 2 days a week, with 48-72 hours between both interventions. Regarding the electrodes, 4 adhesive electrodes (5.0x5.0) will be placed, 2 in the lower lumbar region and two in the parasacral region (S2-S4).

ELIGIBILITY:
Inclusion criteria:

* Adult women
* Pain greater than 3 on the NPRS scale
* Women with regular menstrual cycle, considered regular between 25-30 days

Exclusion criteria:

* Pregnancy or breastfeeding
* Used of intrauterine device
* Diagnosed gynaecological pathology: endometriosis, polycystic ovaries, uterine fibroid, adenomyosis, fibrosis, uterine malformation, pelvic inflammation, scars, SDT...
* Skin lesions that prevent the placement of the electrodes
* Other diagnosed pathologies that contraindicate the application of TENS, neurological pathologies, or cardiovascular diseases
* Absence or doubling of bleeding in one month
* Taking analgesic medications and/or NSAIDs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pain: Numerical Pain Scale (NPRS) | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It evaluates the intensity of menstrual pain in this case. This scale is based on asking the patient about the intensity of their pain between a value of 0, which corresponds to the absence of pain, and a value of 10, which corresponds to the highest possible pain.
Pressure pain threshold (PDU): Analog pressure algometer (Wagner FPX, United States) | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  The subject will be instructed to communicate to the evaluator, as quickly as she perceives the minimum perceptible pain. Measurements were taken in the abdominal area, both on the right and on the left and 4cm from the navel (T10-T12) and in a single point in the lumbar region below the last lumbar vertebra (S2-S4), corresponding to the usual areas of the pain area reported in women with dysmenorrhea. Along with these points, assessments will also be performed bilaterally on the lateral aspect of the arm 10 cm below the lateral border of the acromion (C6-C7), and on the anterior aspect of the thigh 15 cm above the superior of the patella (L2-L3), these latter areas being control areas.
Pain: McGill Pain Index (MPQ) | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  This questionnaire consists of 20 items with the objective of evaluating the different aspects of the patient's perception of pain (sensory perception of pain, emotional affective perception, evaluative perception and the perception of various pains).
Quality of life related to menstruation: Specific quality of life questionnaire related to menstruation (CVM-22) | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It assess the impact of menstruation on the woman's health status during bleeding days. The CVM-22 is a self-administered Likert-type questionnaire, made up of 22 items, where the questionnaire score ranges between 0 and 66, higher scores indicate worse quality of life.
Quality of life: SF12 Health Questionnaire | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It evaluates multidimensional health and it consists of 12 items (physical function, social function, physical role, emotional role, mental health, vitality, body pain and general health). It is a self-administered questionnaire, where the number of response options ranges between 2 and 6, among which the patient can only choose one. This questionnaire allows to obtain two scores, which correspond to the physical summary and the mental summary. A higher score is related to better health status.

SECONDARY OUTCOMES:
Anxiety and Depresion: Hospital Anxiety and Depression Scale (HADS) | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It is a self-administered questionnaire of 14 items, which evaluates anxiety and depression, composed of two subscales of 7 items, one for anxiety (odd items) and another of depression (even items). The intensity or frequency of the symptom is evaluated on a 4-point Likert scale (0-3) with different responses. The time frame, even when the questions are posed in the present, must refer to the previous week.
Catastrophic thinking: Pain Catastrophizing Scale (PCS): | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It is a self-report inventory that assesses pain catastrophizing, composed of 13 items, which are grouped into 3 factors, which are cognitive rumination, magnification, and hopelessness. Using a five-point Likert scale (0, not at all; 1, a little; 2, moderately; 3, a lot; and 4, all the time), the informant rates the intensity with which she has experienced each thought while experiencing pain. The higher the score, the greater the pain catastrophizing, which could be a total of 52 points.
Sleep quality: Pittsburgh Sleep Quality Index (PSQI): | Baseline, immediately after treatment and at 28 days in bleeding phase and sham TENS, while in luteal phase will be done at baseline, at 7 days and at 28 days.
  It is a self-administered questionnaire that measures sleep quality, in addition to the subject's own perception of their sleep. It consists of 24 questions, of which 19 must be answered by the patient themselves (15 closed questions from 0 to 3, and 4 open), while 5 require feedback from the partner or roommate. The 19 self-assessed items are combined to form 7 scoring components (sleep quality, latency, duration, habitual efficiency, sleep disturbances, taking sleep medications, and daytime disturbances), each with a range of 0 to 3. A score of 0 points indicates that there is no difficulty, while a score of 3 corresponds to severe difficulty. The sum of the 7 components would give the global score, which has a range of 0 to 21 points, indicating severe difficulty in all the areas studied, as the score increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Naiara Benítez Aramburu, Torrelavega, Cantabria, Spain

REFERENCES:
- [Result] Iacovides S, Avidon I, Baker FC. What we know about primary dysmenorrhea today: a critical review. Hum Reprod Update. 2015 Nov-Dec;21(6):762-78. doi: 10.1093/humupd/dmv039. Epub 2015 Sep 7. PMID 26346058
- [Result] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Result] ACOG Committee Opinion No. 760: Dysmenorrhea and Endometriosis in the Adolescent. Obstet Gynecol. 2018 Dec;132(6):e249-e258. doi: 10.1097/AOG.0000000000002978. PMID 30461694
- [Result] Coco AS. Primary dysmenorrhea. Am Fam Physician. 1999 Aug;60(2):489-96. PMID 10465224
- [Result] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Result] Osayande AS, Mehulic S. Diagnosis and initial management of dysmenorrhea. Am Fam Physician. 2014 Mar 1;89(5):341-6. PMID 24695505
- [Result] Chen CX, Shieh C, Draucker CB, Carpenter JS. Reasons women do not seek health care for dysmenorrhea. J Clin Nurs. 2018 Jan;27(1-2):e301-e308. doi: 10.1111/jocn.13946. Epub 2017 Sep 7. PMID 28681499
- [Result] Ramos-Pichardo JD, Ortega-Galan AM, Iglesias-Lopez MT, Abreu-Sanchez A, Fernandez-Martinez E. Why Do Some Spanish Nursing Students with Menstrual Pain Fail to Consult Healthcare Professionals? Int J Environ Res Public Health. 2020 Nov 5;17(21):8173. doi: 10.3390/ijerph17218173. PMID 33167417
- [Result] Weissman AM, Hartz AJ, Hansen MD, Johnson SR. The natural history of primary dysmenorrhoea: a longitudinal study. BJOG. 2004 Apr;111(4):345-52. doi: 10.1111/j.1471-0528.2004.00090.x. PMID 15008771
- [Result] Abreu-Sanchez A, Ruiz-Castillo J, Onieva-Zafra MD, Parra-Fernandez ML, Fernandez-Martinez E. Interference and Impact of Dysmenorrhea on the Life of Spanish Nursing Students. Int J Environ Res Public Health. 2020 Sep 5;17(18):6473. doi: 10.3390/ijerph17186473. PMID 32899505
- [Result] Karout S, Soubra L, Rahme D, Karout L, Khojah HMJ, Itani R. Prevalence, risk factors, and management practices of primary dysmenorrhea among young females. BMC Womens Health. 2021 Nov 8;21(1):392. doi: 10.1186/s12905-021-01532-w. PMID 34749716
- [Result] Dawood MY. Primary dysmenorrhea: advances in pathogenesis and management. Obstet Gynecol. 2006 Aug;108(2):428-41. doi: 10.1097/01.AOG.0000230214.26638.0c. PMID 16880317
- [Result] Dawood MY. Dysmenorrhoea and prostaglandins: pharmacological and therapeutic considerations. Drugs. 1981 Jul;22(1):42-56. doi: 10.2165/00003495-198122010-00003. PMID 6790261
- [Result] PICKLES VR. Myometrial responses to the menstrual plain muscle stimulant. J Endocrinol. 1959 Nov;19:150-7. doi: 10.1677/joe.0.0190150. No abstract available. PMID 14432762
- [Result] Maybin JA, Critchley HO. Menstrual physiology: implications for endometrial pathology and beyond. Hum Reprod Update. 2015 Nov-Dec;21(6):748-61. doi: 10.1093/humupd/dmv038. Epub 2015 Aug 7. PMID 26253932
- [Result] Messing K, Saurel-Cubizolles MJ, Bourgine M, Kaminski M. Factors associated with dysmenorrhea among workers in French poultry slaughterhouses and canneries. J Occup Med. 1993 May;35(5):493-500. PMID 8515321
- [Result] Sundell G, Milsom I, Andersch B. Factors influencing the prevalence and severity of dysmenorrhoea in young women. Br J Obstet Gynaecol. 1990 Jul;97(7):588-94. doi: 10.1111/j.1471-0528.1990.tb02545.x. PMID 2390501
- [Result] Harlow SD, Park M. A longitudinal study of risk factors for the occurrence, duration and severity of menstrual cramps in a cohort of college women. Br J Obstet Gynaecol. 1996 Nov;103(11):1134-42. doi: 10.1111/j.1471-0528.1996.tb09597.x. PMID 8917003
- [Result] Hu Z, Tang L, Chen L, Kaminga AC, Xu H. Prevalence and Risk Factors Associated with Primary Dysmenorrhea among Chinese Female University Students: A Cross-sectional Study. J Pediatr Adolesc Gynecol. 2020 Feb;33(1):15-22. doi: 10.1016/j.jpag.2019.09.004. Epub 2019 Sep 17. PMID 31539615
- [Result] Thorbert G, Alm P, Owman C, Sjoberg NO, Sporrong B. Regional changes in structural and functional integrity of myometrial adrenergic nerves in pregnant guinea-pig, and their relationship to the localization of the conceptus. Acta Physiol Scand. 1978 Jun;103(2):120-31. doi: 10.1111/j.1748-1716.1978.tb06199.x. PMID 676764
- [Result] Montero P, Bernis C, Fernandez V, Castro S. Influence of body mass index and slimming habits on menstrual pain and cycle irregularity. J Biosoc Sci. 1996 Jul;28(3):315-23. doi: 10.1017/s0021932000022380. PMID 8698711
- [Result] Parazzini F, Tozzi L, Mezzopane R, Luchini L, Marchini M, Fedele L. Cigarette smoking, alcohol consumption, and risk of primary dysmenorrhea. Epidemiology. 1994 Jul;5(4):469-72. doi: 10.1097/00001648-199407000-00016. PMID 7918820
- [Result] Burnett M, Lemyre M. No. 345-Primary Dysmenorrhea Consensus Guideline. J Obstet Gynaecol Can. 2017 Jul;39(7):585-595. doi: 10.1016/j.jogc.2016.12.023. PMID 28625286
- [Result] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Result] Campbell MA, McGrath PJ. Use of medication by adolescents for the management of menstrual discomfort. Arch Pediatr Adolesc Med. 1997 Sep;151(9):905-13. doi: 10.1001/archpedi.1997.02170460043007. PMID 9308868
- [Result] Dawood MY. Nonsteroidal anti-inflammatory drugs and changing attitudes toward dysmenorrhea. Am J Med. 1988 May 20;84(5A):23-9. doi: 10.1016/0002-9343(88)90473-1. PMID 3287908
- [Result] Parra-Fernandez ML, Onieva-Zafra MD, Abreu-Sanchez A, Ramos-Pichardo JD, Iglesias-Lopez MT, Fernandez-Martinez E. Management of Primary Dysmenorrhea among University Students in the South of Spain and Family Influence. Int J Environ Res Public Health. 2020 Aug 1;17(15):5570. doi: 10.3390/ijerph17155570. PMID 32752254
- [Result] Dmitrovic R, Kunselman AR, Legro RS. Continuous compared with cyclic oral contraceptives for the treatment of primary dysmenorrhea: a randomized controlled trial. Obstet Gynecol. 2012 Jun;119(6):1143-50. doi: 10.1097/AOG.0b013e318257217a. PMID 22617578
- [Result] Edelman A, Micks E, Gallo MF, Jensen JT, Grimes DA. Continuous or extended cycle vs. cyclic use of combined hormonal contraceptives for contraception. Cochrane Database Syst Rev. 2014 Jul 29;2014(7):CD004695. doi: 10.1002/14651858.CD004695.pub3. PMID 25072731
- [Result] Milsom I, Hedner N, Mannheimer C. A comparative study of the effect of high-intensity transcutaneous nerve stimulation and oral naproxen on intrauterine pressure and menstrual pain in patients with primary dysmenorrhea. Am J Obstet Gynecol. 1994 Jan;170(1 Pt 1):123-9. doi: 10.1016/s0002-9378(94)70396-5. PMID 8296814
- [Result] Ruoff G, Lema M. Strategies in pain management: new and potential indications for COX-2 specific inhibitors. J Pain Symptom Manage. 2003 Feb;25(2 Suppl):S21-31. doi: 10.1016/s0885-3924(02)00628-0. PMID 12604154
- [Result] Di Girolamo G, Sanchez AJ, De Los Santos AR, Gonzalez CD. Is acetaminophen, and its combination with pamabrom, an effective therapeutic option in primary dysmenorrhoea? Expert Opin Pharmacother. 2004 Mar;5(3):561-70. doi: 10.1517/14656566.5.3.561. PMID 15013925
- [Result] Abubakar U, Zulkarnain AI, Samri F, Hisham SR, Alias A, Ishak M, Sugiman H, Ghozali T. Use of complementary and alternative therapies for the treatment of dysmenorrhea among undergraduate pharmacy students in Malaysia: a cross sectional study. BMC Complement Med Ther. 2020 Sep 18;20(1):285. doi: 10.1186/s12906-020-03082-4. PMID 32948163
- [Result] Akin MD, Weingand KW, Hengehold DA, Goodale MB, Hinkle RT, Smith RP. Continuous low-level topical heat in the treatment of dysmenorrhea. Obstet Gynecol. 2001 Mar;97(3):343-9. doi: 10.1016/s0029-7844(00)01163-7. PMID 11239634
- [Result] Armour M, Smith CA, Steel KA, Macmillan F. The effectiveness of self-care and lifestyle interventions in primary dysmenorrhea: a systematic review and meta-analysis. BMC Complement Altern Med. 2019 Jan 17;19(1):22. doi: 10.1186/s12906-019-2433-8. PMID 30654775
- [Result] Armour M, Ee CC, Naidoo D, Ayati Z, Chalmers KJ, Steel KA, de Manincor MJ, Delshad E. Exercise for dysmenorrhoea. Cochrane Database Syst Rev. 2019 Sep 20;9(9):CD004142. doi: 10.1002/14651858.CD004142.pub4. PMID 31538328
- [Result] Tsonis O, Gkrozou F, Barmpalia Z, Makopoulou A, Siafaka V. Integrating Lifestyle Focused Approaches into the Management of Primary Dysmenorrhea: Impact on Quality of Life. Int J Womens Health. 2021 Mar 17;13:327-336. doi: 10.2147/IJWH.S264023. eCollection 2021. PMID 33762855
- [Result] Jaleel G, Shaphe MA, Khan AR, Malhotra D, Khan H, Parveen S, Qasheesh M, Beg RA, Chahal A, Ahmad F, Ahmad MF. Effect of Exercises on Central and Endocrine System for Pain Modulation in Primary Dysmenorrhea. J Lifestyle Med. 2022 Jan 31;12(1):15-25. doi: 10.15280/jlm.2022.12.1.15. PMID 35300040
- [Result] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122
- [Result] Ortiz MI, Cortes-Marquez SK, Romero-Quezada LC, Murguia-Canovas G, Jaramillo-Diaz AP. Effect of a physiotherapy program in women with primary dysmenorrhea. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:24-9. doi: 10.1016/j.ejogrb.2015.08.008. Epub 2015 Aug 17. PMID 26319652
- [Result] Azima S, Bakhshayesh HR, Kaviani M, Abbasnia K, Sayadi M. Comparison of the Effect of Massage Therapy and Isometric Exercises on Primary Dysmenorrhea: A Randomized Controlled Clinical Trial. J Pediatr Adolesc Gynecol. 2015 Dec;28(6):486-91. doi: 10.1016/j.jpag.2015.02.003. Epub 2015 Mar 5. PMID 26272447
- [Result] Gaubeca-Gilarranz A, Fernandez-de-Las-Penas C, Medina-Torres JR, Seoane-Ruiz JM, Company-Palones A, Cleland JA, Arias-Buria JL. Effectiveness of dry needling of rectus abdominis trigger points for the treatment of primary dysmenorrhoea: a randomised parallel-group trial. Acupunct Med. 2018 Oct;36(5):302-310. doi: 10.1136/acupmed-2017-011566. Epub 2018 May 2. PMID 29720379
- [Result] Smith CA, Armour M, Zhu X, Li X, Lu ZY, Song J. Acupuncture for dysmenorrhoea. Cochrane Database Syst Rev. 2016 Apr 18;4(4):CD007854. doi: 10.1002/14651858.CD007854.pub3. PMID 27087494
- [Result] Sharghi M, Mansurkhani SM, Larky DA, Kooti W, Niksefat M, Firoozbakht M, Behzadifar M, Azami M, Servatyari K, Jouybari L. An update and systematic review on the treatment of primary dysmenorrhea. JBRA Assist Reprod. 2019 Jan 31;23(1):51-57. doi: 10.5935/1518-0557.20180083. PMID 30521155
- [Result] Abaraogu UO, Igwe SE, Tabansi-Ochiogu CS, Duru DO. A Systematic Review and Meta-Analysis of the Efficacy of Manipulative Therapy in Women with Primary Dysmenorrhea. Explore (NY). 2017 Nov-Dec;13(6):386-392. doi: 10.1016/j.explore.2017.08.001. Epub 2017 Aug 30. PMID 28988817
- [Result] Dogan H, Eroglu S, Akbayrak T. The effect of kinesio taping and lifestyle changes on pain, body awareness and quality of life in primary dysmenorrhea. Complement Ther Clin Pract. 2020 May;39:101120. doi: 10.1016/j.ctcp.2020.101120. Epub 2020 Feb 22. PMID 32379659
- [Result] Apay SE, Arslan S, Akpinar RB, Celebioglu A. Effect of aromatherapy massage on dysmenorrhea in Turkish students. Pain Manag Nurs. 2012 Dec;13(4):236-40. doi: 10.1016/j.pmn.2010.04.002. Epub 2010 Sep 15. PMID 23158705
- [Result] Lee MS, Lee HW, Khalil M, Lim HS, Lim HJ. Aromatherapy for Managing Pain in Primary Dysmenorrhea: A Systematic Review of Randomized Placebo-Controlled Trials. J Clin Med. 2018 Nov 10;7(11):434. doi: 10.3390/jcm7110434. PMID 30423839
- [Result] Lauretti GR, Oliveira R, Parada F, Mattos AL. The New Portable Transcutaneous Electrical Nerve Stimulation Device Was Efficacious in the Control of Primary Dysmenorrhea Cramp Pain. Neuromodulation. 2015 Aug;18(6):522-6; discussion 522-7. doi: 10.1111/ner.12269. Epub 2015 Feb 5. PMID 25655828
- [Result] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Result] Treede RD. Gain control mechanisms in the nociceptive system. Pain. 2016 Jun;157(6):1199-1204. doi: 10.1097/j.pain.0000000000000499. PMID 26817644
- [Result] Mayer DJ, Hayes RL. Stimulation-produced analgesia: development of tolerance and cross-tolerance to morphine. Science. 1975 May 30;188(4191):941-3. doi: 10.1126/science.1094537.
- [Result] Petrovic P, Kalso E, Petersson KM, Ingvar M. Placebo and opioid analgesia-- imaging a shared neuronal network. Science. 2002 Mar 1;295(5560):1737-40. doi: 10.1126/science.1067176. Epub 2002 Feb 7. PMID 11834781
- [Result] Wang SF, Lee JP, Hwa HL. Effect of transcutaneous electrical nerve stimulation on primary dysmenorrhea. Neuromodulation. 2009 Oct;12(4):302-9. doi: 10.1111/j.1525-1403.2009.00226.x. Epub 2009 Aug 20. PMID 22151421
- [Result] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- [Result] Budgell BS, Sovak G, Soave D. TENS augments blood flow in somatotopically linked spinal cord segments and mitigates compressive ischemia. Spinal Cord. 2014 Oct;52(10):744-8. doi: 10.1038/sc.2014.120. Epub 2014 Jul 22. PMID 25047054
- [Result] Dawood MY, Ramos J. Transcutaneous electrical nerve stimulation (TENS) for the treatment of primary dysmenorrhea: a randomized crossover comparison with placebo TENS and ibuprofen. Obstet Gynecol. 1990 Apr;75(4):656-60. PMID 2179780
- [Result] Lewers D, Clelland JA, Jackson JR, Varner RE, Bergman J. Transcutaneous electrical nerve stimulation in the relief of primary dysmenorrhea. Phys Ther. 1989 Jan;69(1):3-9. doi: 10.1093/ptj/69.1.3. PMID 2783493
- [Result] Elboim-Gabyzon M, Kalichman L. Transcutaneous Electrical Nerve Stimulation (TENS) for Primary Dysmenorrhea: An Overview. Int J Womens Health. 2020 Jan 8;12:1-10. doi: 10.2147/IJWH.S220523. eCollection 2020. PMID 32021488
- [Result] Proctor ML, Smith CA, Farquhar CM, Stones RW. Transcutaneous electrical nerve stimulation and acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2002;2002(1):CD002123. doi: 10.1002/14651858.CD002123. PMID 11869624
- [Result] Bai HY, Bai HY, Yang ZQ. Effect of transcutaneous electrical nerve stimulation therapy for the treatment of primary dysmenorrheal. Medicine (Baltimore). 2017 Sep;96(36):e7959. doi: 10.1097/MD.0000000000007959. PMID 28885348
- [Result] Bergeron-Vezina K, Leonard G. On "what makes transcutaneous electrical nerve stimulation work?..." Sluka KA, Bjordal JM, Marchand S, Rakel BA. Phys Ther. 2013;93:1397-1402. Phys Ther. 2013 Oct;93(10):1426-7. doi: 10.2522/ptj.2013.93.10.1426. No abstract available. PMID 24086069
- [Result] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Result] Reading AE. The internal structure of the McGill pain questionnaire in dysmenorrhoea patients. Pain. 1979 Dec;7(3):353-358. doi: 10.1016/0304-3959(79)90091-5. PMID 530741
- [Result] Lazaro C, Caseras X, Whizar-Lugo VM, Wenk R, Baldioceda F, Bernal R, Ovalle A, Torrubia R, Banos JE. Psychometric properties of a Spanish version of the McGill Pain Questionnaire in several Spanish-speaking countries. Clin J Pain. 2001 Dec;17(4):365-74. doi: 10.1097/00002508-200112000-00012. PMID 11783818
- [Result] Masedo AI, Esteve R. Some empirical evidence regarding the validity of the Spanish version of the McGill Pain Questionnaire (MPQ-SV). Pain. 2000 Apr;85(3):451-456. doi: 10.1016/S0304-3959(99)00300-0. PMID 10781918
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Result] Monteagudo Piqueras O, Hernando Arizaleta L, Palomar Rodriguez JA. [Population based norms of the Spanish version of the SF-12V2 for Murcia (Spain)]. Gac Sanit. 2011 Jan-Feb;25(1):50-61. doi: 10.1016/j.gaceta.2010.09.001. Epub 2010 Oct 25. Spanish. PMID 20980078
- [Result] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Result] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Result] Morris JL, Rohay J, Chasens ER. Sex Differences in the Psychometric Properties of the Pittsburgh Sleep Quality Index. J Womens Health (Larchmt). 2018 Mar;27(3):278-282. doi: 10.1089/jwh.2017.6447. Epub 2017 Nov 20. PMID 29154713
- [Result] Beck SL, Schwartz AL, Towsley G, Dudley W, Barsevick A. Psychometric evaluation of the Pittsburgh Sleep Quality Index in cancer patients. J Pain Symptom Manage. 2004 Feb;27(2):140-8. doi: 10.1016/j.jpainsymman.2003.12.002. PMID 15157038
- [Result] Bisset LM, Evans K, Tuttle N. Reliability of 2 protocols for assessing pressure pain threshold in healthy young adults. J Manipulative Physiol Ther. 2015 May;38(4):282-7. doi: 10.1016/j.jmpt.2015.03.001. Epub 2015 Apr 27. PMID 25925018
- [Result] Fischer AA. Pressure algometry over normal muscles. Standard values, validity and reproducibility of pressure threshold. Pain. 1987 Jul;30(1):115-126. doi: 10.1016/0304-3959(87)90089-3. PMID 3614975
- [Result] Nie H, Arendt-Nielsen L, Andersen H, Graven-Nielsen T. Temporal summation of pain evoked by mechanical stimulation in deep and superficial tissue. J Pain. 2005 Jun;6(6):348-55. doi: 10.1016/j.jpain.2005.01.352. PMID 15943956
- [Result] Bajaj P, Bajaj P, Madsen H, Arendt-Nielsen L. A comparison of modality-specific somatosensory changes during menstruation in dysmenorrheic and nondysmenorrheic women. Clin J Pain. 2002 May-Jun;18(3):180-90. doi: 10.1097/00002508-200205000-00007. PMID 12048420
- [Result] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Result] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Result] Reed BG, Carr BR. The Normal Menstrual Cycle and the Control of Ovulation. 2018 Aug 5. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279054/ PMID 25905282
- [Result] Hampson E. A brief guide to the menstrual cycle and oral contraceptive use for researchers in behavioral endocrinology. Horm Behav. 2020 Mar;119:104655. doi: 10.1016/j.yhbeh.2019.104655. Epub 2019 Dec 23. PMID 31843564
- [Result] Mihm M, Gangooly S, Muttukrishna S. The normal menstrual cycle in women. Anim Reprod Sci. 2011 Apr;124(3-4):229-36. doi: 10.1016/j.anireprosci.2010.08.030. Epub 2010 Sep 3. PMID 20869180
- [Result] Rodrigues JC, Avila MA, Driusso P. Transcutaneous electrical nerve stimulation for women with primary dysmenorrhea: Study protocol for a randomized controlled clinical trial with economic evaluation. PLoS One. 2021 May 20;16(5):e0250111. doi: 10.1371/journal.pone.0250111. eCollection 2021. PMID 34014922
- [Result] Machado AFP, Perracini MR, Rampazo EP, Driusso P, Liebano RE. Effects of thermotherapy and transcutaneous electrical nerve stimulation on patients with primary dysmenorrhea: A randomized, placebo-controlled, double-blind clinical trial. Complement Ther Med. 2019 Dec;47:102188. doi: 10.1016/j.ctim.2019.08.022. Epub 2019 Aug 28. PMID 31779988
- [Result] Yokozuka M, Nagai M, Katsura R, Kenmyo K. Analgesia by Sacral Surface Electrical Stimulation for Primary Dysmenorrhoea. J Rehabil Med Clin Commun. 2020 Feb 27;3:1000027. doi: 10.2340/20030711-1000027. eCollection 2020. PMID 33884129